CLINICAL TRIAL: NCT02679079
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Assess the Safety and Efficacy of NBI-98854 in Pediatric Subjects With Tourette Syndrome
Brief Title: Safety and Efficacy Study of NBI-98854 in Children and Adolescents With Tourette Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neurocrine Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NBI-98854-1501
Record Dates: First submitted 2016-02-05; First posted 2016-02-10 (Estimated); Results first posted 2021-01-15 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2020-12

CONDITIONS: Tourette Syndrome
MeSH Terms: conditions — Tourette Syndrome | interventions — valbenazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Administered once daily for 6 weeks
  Interventions: Drug: Placebo
- Dose Group 1 (Experimental): Administered once daily for 6 weeks
  Interventions: Drug: NBI-98854
- Dose Group 2 (Experimental): Administered once daily for 6 weeks
  Interventions: Drug: NBI-98854

INTERVENTIONS:
Drug: NBI-98854
  Arms: Dose Group 1; Dose Group 2
Drug: Placebo
  Arms: Placebo

SUMMARY:
Phase 2, double-blind, placebo-controlled study to assess the safety and efficacy of NBI-98854 administered once daily (qd) for a total of 6 weeks of treatment. This study will enroll approximately 90 male and female pediatric subjects clinically diagnosed with Tourette Syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. Have a clinical diagnosis of Tourette Syndrome (TS)
2. Have at least moderate tic severity
3. Have TS symptoms that impair school, occupational, and/or social function
4. If using maintenance medication(s) for TS or TS spectrum diagnoses (e.g. obsessive-compulsive disorder [OCD], Attention-Deficit Hyperactivity Disorder [ADHD]), be on stable doses
5. Be in good general health
6. Adolescent subjects (12 to 17 years of age) must have a negative urine drug screen for amphetamines, barbiturates, benzodiazepine, phencyclidine, cocaine, opiates, or cannabinoids and a negative alcohol screen
7. Subjects of childbearing potential who do not practice total abstinence must agree to use hormonal or two forms of nonhormonal contraception (dual contraception) consistently during the screening, treatment and follow-up periods of the study

Exclusion Criteria:

1. Have an active, clinically significant unstable medical condition within 1 month prior to screening
2. Have a known history of long QT syndrome or cardiac arrhythmia
3. Have a known history of neuroleptic malignant syndrome
4. Have a cancer diagnosis within 3 years prior to screening (some exceptions allowed)
5. Have an allergy, hypersensitivity, or intolerance to VMAT2 inhibitors
6. Have a blood loss ≥250 mL or donated blood within 30 days prior to screening
7. Have a known history of substance dependence, substance (drug) or alcohol abuse
8. Have a significant risk of suicidal or violent behavior
9. Have initiated Comprehensive Behavioral Intervention for Tics (CBIT) during the screening period or at baseline or plan to initiate CBIT during the study
10. Have received an investigational drug within 30 days before screening or plan to use an investigational drug (other than NBI-98854) during the study

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 98 (Actual)
Dates: Start 2016-03-23 (Actual); Primary Completion 2017-04-14 (Actual); Study Completion 2017-04-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (44):
- United States (44):
  - Sun City, Arizona
  - Springdale, Arkansas
  - Long Beach, California
  - San Bernardino, California
  - San Diego, California
  - Upland, California
  - Bradenton, Florida
  - Gainesville, Florida
  - Hialeah, Florida
  - Loxahatchee Groves, Florida
  - Melbourne, Florida
  - Orlando, Florida
  - St. Petersburg, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Naperville, Illinois
  - Wichita, Kansas
  - Boston, Massachusetts
  - Natick, Massachusetts
  - Ann Arbor, Michigan
  - Bloomfield Hills, Michigan
  - Lincoln, Nebraska
  - Nashua, New Hampshire
  - Marlton, New Jersey
  - Summit, New Jersey
  - Manhasset, New York
  - New York, New York
  - Rochester, New York
  - Cincinnati, Ohio
  - Middleburg Heights, Ohio
  - Oklahoma City, Oklahoma
  - Franklin, Tennessee
  - Nashville, Tennessee
  - Dallas, Texas
  - DeSoto, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - Irving, Texas
  - Orem, Utah
  - Salt Lake City, Utah
  - Kirkland, Washington
  - Seattle, Washington
  - Spokane, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled participants (male and female), 6 to 17 years of age, with a diagnosis of Tourette Syndrome through Diagnostic and Statistical Manual of Mental Disorders, 4th or 5th Editions (DSM-IV or -V) from 30 study centers in the United States. The first participant was enrolled on 23 March 2016 and last participant completed the study on 14 April 2017.
Groups:
- Placebo: Participants received matching placebo once daily for 6 weeks.
- NBI-98854 Low Dose: Participants received valbenazine once daily for 6 weeks. Participants aged 6 to 11 years received 10 mg/day. Participants aged 12 to 17 years received 20 mg/day.
- NBI-98854 High Dose: Participants received valbenazine once daily for 6 weeks. Participants aged 6 to 11 years received 10 mg/day for the first week followed by 20 mg/day for the remainder of the treatment period. Participants aged 12 to 17 years received 20 mg/day for the first week followed by 40 mg/day for the remainder of the treatment period.
Period: Overall Study
Arm/Group | Placebo | NBI-98854 Low Dose | NBI-98854 High Dose
Started | 33 | 32 | 33
ITT Analysis Set (Intent-to-treat (ITT) analysis set included all randomized participants who received at least one dose of study drug, had postbaseline safety data, and had a baseline (Day -1) and at least one postrandomization Total Tic Score (TTS) value reported at a scheduled or mapped early termination (ET) visit during the 6 week treatment period.) | 31 | 32 | 32
Completed | 29 | 30 | 31
Not Completed | 4 | 2 | 2
Not completed — Adverse Event | 2 | 0 | 2
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) analysis set included all randomized participants who received at least one dose of study drug, had postbaseline safety data, and had a baseline (Day -1) and at least one postrandomization Total Tic Score (TTS) value reported at a scheduled or mapped early termination (ET) visit during the 6 week treatment period.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | NBI-98854 Low Dose | NBI-98854 High Dose | Total
Number analyzed (Participants) | 31 | 32 | 32 | 95
Age, Continuous [Mean (Full Range); unit: Years] | 11.5 [7 to 15] | 12.0 [6 to 17] | 11.6 [6 to 17] | 11.7 [6 to 17]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 11 | 5 | 20
  Male | 27 | 21 | 27 | 75
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 4 | 2 | 11
  Not Hispanic or Latino | 26 | 28 | 30 | 84
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 2 | 5
  White | 27 | 31 | 29 | 87
  More than one race | 2 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0
Yale Global Tic Severity Scale (YGTSS) Total Tic Score (TTS) [Mean (Full Range); unit: Score on scale] — The YGTSS is designed to rate the overall severity of motor and phonic tic symptoms across a range of dimensions: number, frequency, intensity, complexity, and interference. The YGTSS was administered by the investigator (or qualified designee) using a computer-based structured clinical interview. The TTS is the sum of the 5 motor tic items and the 5 phonic (vocal) tic items and ranges from 0 to 50, with higher scores representing greater severity
  Score on scale | 30.4 [9 to 44] | 32.8 [23 to 49] | 32.9 [24 to 47] | 32.1 [9 to 49]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 6 in the Yale Global Tic Severity Scale (YGTSS) Total Tic Score (TTS)
Description: The YGTSS is designed to rate the overall severity of motor and phonic tic symptoms across a range of dimensions: number, frequency, intensity, complexity, and interference. The YGTSS was administered by the investigator (or qualified designee) using a computer-based structured clinical interview. The TTS is the sum of the 5 motor tic items and the 5 phonic (vocal) tic items and ranges from 0 to 50, with higher scores representing greater severity
Time Frame: Baseline, Week 6
Population: The intent-to-treat (ITT) analysis set included all randomized participants who received at least one dose of study drug, had postbaseline safety data, and had a baseline (Day -1) and at least one postrandomization TTS value reported at a scheduled or mapped early termination (ET) visit during the 6-week treatment period. Dose levels based on age group were prespecified to be combined within each dose arm.
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Placebo | NBI-98854 Low Dose | NBI-98854 High Dose
Number analyzed (Participants) | 31 | 32 | 32
Score on scale | -8.8 (1.5) | -7.3 (1.4) | -9.1 (1.4)
Statistical Analysis 1: Comparison: Placebo vs NBI-98854 High Dose; Test type: Superiority; p = 0.89, Mixed Models Analysis — Nominal p-value is considered statistically significant if less than 0.05. To control for multiplicity, comparisons were tested sequentially; Mean Difference (Net) = -0.3, 95% CI 2-sided [-4.4 to 3.8], Standard Error of Mean 2.1
Statistical Analysis 2: Comparison: Placebo vs NBI-98854 Low Dose; Test type: Superiority; p = 0.47, Mixed Models Analysis — To control for multiplicity, comparisons were tested sequentially. Nominal p-value was not evaluated for statistical significance since first comparison was not statistically significant; Mean Difference (Net) = 1.5, 95% CI 2-sided [-2.6 to 5.6], Standard Error of Mean 2.1

2. Secondary Outcome: Clinical Global Impression of Tourette Syndrome (CGI-TS) - Improvement Score at Week 6
Description: The CGI-TS-Improvement scale is used to assess overall improvement since the initiation of study drug dosing on a 7-point scale. Each of the CGI-TS-Improvement response categories was assigned a numerical score as follows: 1 = Very much improved; 2 = Much improved; 3 = Minimally improved; 4 = Not changed; 5 = Minimally worse; 6 = Much worse; 7 = Very much worse.
Time Frame: Week 6
Population: The ITT analysis set included all randomized participants who received at least one dose of study drug, had postbaseline safety data, and had a baseline (Day -1) and at least one postrandomization TTS value reported at a scheduled or mapped early termination (ET) visit during the 6-week treatment period. Dose levels based on age group were prespecified to be combined within each dose arm.
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Placebo | NBI-98854 Low Dose | NBI-98854 High Dose
Number analyzed (Participants) | 31 | 32 | 32
Score on scale | 3.4 (0.2) | 3.5 (0.2) | 3.0 (0.2)
Statistical Analysis 1: Comparison: Placebo vs NBI-98854 High Dose; Test type: Superiority; p = 0.21, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Net) = -0.4, 95% CI 2-sided [-1.0 to 0.2], Standard Error of Mean 0.3
Statistical Analysis 2: Comparison: Placebo vs NBI-98854 Low Dose; Test type: Superiority; p = 0.67, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Net) = 0.1, 95% CI 2-sided [-0.5 to 0.8], Standard Error of Mean 0.3

3. Secondary Outcome: Participants Who Are a YGTSS TTS Responder at Week 6
Description: A TTS responder is defined, on a per-visit basis, as a participant whose TTS value is reduced by at least 30% from baseline at the specified postbaseline visit.
Time Frame: Baseline, Week 6
Population: Participants with observed data in the ITT analysis set, defined as all randomized participants who received at least one dose of study drug, had postbaseline safety data, and had a baseline (Day -1) and at least one postrandomization TTS value reported at a scheduled or mapped early termination (ET) visit during the 6-week treatment period. Dose levels based on age group were prespecified to be combined within each dose arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | NBI-98854 Low Dose | NBI-98854 High Dose
Number analyzed (Participants) | 29 | 30 | 31
Participants | 10 | 9 | 15
Statistical Analysis 1: Comparison: Placebo vs NBI-98854 High Dose; Test type: Superiority; p = 0.24, Cochran-Mantel-Haenszel — Comparison was not included in multiplicity adjustment procedure; Stratified by age group (6 to 11 years, 12 to 17 years); Risk Difference (RD) = 13.9 — Risk difference expressed as percentage
Statistical Analysis 2: Comparison: Placebo vs NBI-98854 Low Dose; Test type: Superiority; p = 0.71, Cochran-Mantel-Haenszel — Comparison was not included in multiplicity adjustment procedure; Stratified by age group (6 to 11 years, 12 to 17 years); Risk Difference (RD) = -4.5 — Risk difference expressed as a percentage

4. Secondary Outcome: Change From Baseline to Week 6 in the YGTSS Impairment Score
Description: The YGTSS Impairment item is used to rate impairment due to tics using the following 50-point anchored scale: 0 = None; 10 = Minimal; 20 = Mild; 30 = Moderate; 40 = Marked; 50 = Severe.
Time Frame: Baseline, Week 6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Placebo | NBI-98854 Low Dose | NBI-98854 High Dose
Number analyzed (Participants) | 31 | 32 | 32
Score on scale | -8.5 (2.1) | -7.1 (2.1) | -10.4 (2.0)
Statistical Analysis 1: Comparison: Placebo vs NBI-98854 High Dose; Test type: Superiority; p = 0.52, Mixed Models Analysis — Comparison was not included in multiplicity adjustment procedure; Mean Difference (Net) = -1.9, 95% CI 2-sided [-7.7 to 3.9], Standard Error of Mean 2.9
Statistical Analysis 2: Comparison: Placebo vs NBI-98854 Low Dose; Test type: Superiority; p = 0.64, Mixed Models Analysis — Comparison was not included in multiplicity adjustment procedure; Mean Difference (Net) = 1.4, 95% CI 2-sided [-4.5 to 7.2], Standard Error of Mean 2.9

5. Secondary Outcome: Change From Baseline to Week 6 in the YGTSS Global Tic Severity Score
Description: The YGTSS Global Tic Severity score is the sum of the YGTSS TTS and the YGTSS Impairment score and ranges from 0 to 100, with higher scores representing greater severity.
Time Frame: Baseline, Week 6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Placebo | NBI-98854 Low Dose | NBI-98854 High Dose
Number analyzed (Participants) | 31 | 32 | 32
Score on scale | -17.2 (3.2) | -14.4 (3.1) | -19.5 (3.1)
Statistical Analysis 1: Comparison: Placebo vs NBI-98854 High Dose; Test type: Superiority; p = 0.60, Mixed Models Analysis — Comparison was not included in multiplicity adjustment procedure; Mean Difference (Net) = -2.3, 95% CI 2-sided [-11.2 to 6.5], Standard Error of Mean 4.5
Statistical Analysis 2: Comparison: Placebo vs NBI-98854 Low Dose; Test type: Superiority; p = 0.54, Mixed Models Analysis — Comparison was not included in multiplicity adjustment procedure; Mean Difference (Net) = 2.8, 95% CI 2-sided [-6.1 to 11.7], Standard Error of Mean 4.5

6. Secondary Outcome: Change From Baseline to Week 6 in the Rush Video-based Tic Rating Scale (RTRS) Total Score
Description: A modified RTRS was used in this study that includes short video recordings to measure 5 tic variables: number of body areas affected, frequency of motor and phonic tics, and severity of motor and phonic tics. The RTRS total score is calculated as the sum of the 5 domain scores, and ranges from 0 to 20, with higher scores representing greater severity. The final on-treatment visit was used in participants who discontinued prior to Week 6.
Time Frame: Baseline, Week 6
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Placebo | NBI-98854 Low Dose | NBI-98854 High Dose
Number analyzed (Participants) | 28 | 27 | 30
Score on scale | -1.2 (0.8) | -1.6 (0.8) | -1.7 (0.7)
Statistical Analysis 1: Comparison: Placebo vs NBI-98854 High Dose; Test type: Superiority; p = 0.64, ANCOVA — Comparison was not included in multiplicity adjustment procedure; Mean Difference (Net) = -0.5, 95% CI 2-sided [-2.6 to 1.6], Standard Error of Mean 1.1
Statistical Analysis 2: Comparison: Placebo vs NBI-98854 Low Dose; Test type: Superiority; p = 0.77, ANCOVA — Comparison was not included in multiplicity adjustment procedure; Mean Difference (Net) = -0.3, 95% CI 2-sided [-2.5 to 1.9], Standard Error of Mean 1.1

7. Secondary Outcome: Change From Baseline to Week 6 in the Premonitory Urge for Tics Scale (PUTS) Total Score
Description: The PUTS is an instrument for quantifying the premonitory urge phenomena associated with tics. It consists of 9 items, each of which is scored on a 4-point scale (1=not at all true, 2=a little true, 3=pretty much true, 4=very much true). The PUTS total score is calculated as the sum of the scores for the 9 items. The total score ranges from 9 to 36, with higher scores indicating a worse outcome.
Time Frame: Baseline, Week 6
Population: The ITT analysis set included all randomized participants who received at least one dose of study drug, had postbaseline safety data, and had a baseline (Day -1) and at least one postrandomization TTS value reported at a scheduled or mapped early termination (ET) visit during the 6-week treatment period. Excludes those with missing PUTS data. Dose levels based on age group were prespecified to be combined within each dose arm.
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Placebo | NBI-98854 Low Dose | NBI-98854 High Dose
Number analyzed (Participants) | 31 | 32 | 31
Score on scale | -0.6 (0.8) | -1.0 (0.8) | 0.3 (0.8)
Statistical Analysis 1: Comparison: Placebo vs NBI-98854 High Dose; Test type: Superiority; p = 0.45, Mixed Models Analysis — Comparison was not included in multiplicity adjustment procedure; Mean Difference (Net) = 0.9, 95% CI 2-sided [-1.4 to 3.2], Standard Error of Mean 1.2
Statistical Analysis 2: Comparison: Placebo vs NBI-98854 Low Dose; Test type: Superiority; p = 0.72, Mixed Models Analysis — Comparison was not included in multiplicity adjustment procedure; Mean Difference (Net) = -0.4, 95% CI 2-sided [-2.7 to 1.9], Standard Error of Mean 1.2

8. Secondary Outcome: Change From Baseline to Week 6 in the Clinical Global Impression of Tics (CGI-Tics) - Severity Score
Description: The CGI-Tics-Severity scale is used to assess overall severity on a 7-point scale. Each of the CGI-Tics-Severity response categories was assigned a numerical score as follows: 1 = Normal, not at all ill; 2 = Borderline ill; 3 = Mildly ill; 4 = Moderately ill; 5 = Markedly ill; 6 = Severely ill; 7 = Among the most extremely ill patient.
Time Frame: Baseline, Week 6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Placebo | NBI-98854 Low Dose | NBI-98854 High Dose
Number analyzed (Participants) | 31 | 32 | 32
Score on scale | -1.1 (0.2) | -0.5 (0.2) | -0.9 (0.2)
Statistical Analysis 1: Comparison: Placebo vs NBI-98854 High Dose; Test type: Superiority; p = 0.41, Mixed Models Analysis — Comparison was not included in multiplicity adjustment procedure; Mean Difference (Net) = 0.2, 95% CI 2-sided [-0.3 to 0.7], Standard Error of Mean 0.2
Statistical Analysis 2: Comparison: Placebo; Test type: Superiority; p = 0.01, Mixed Models Analysis — Comparison was not included in multiplicity adjustment procedure; Mean Difference (Net) = 0.6, 95% CI 2-sided [0.2 to 1.1], Standard Error of Mean 0.2

9. Secondary Outcome: Participants Who Are a CGI-TS-Improvement Responder at Week 6
Description: A participant is classified as a CGI-TS-Improvement responder at a given visit if their CGI-TS-Improvement score is either a "1" ("very much improved") or a "2" ("much improved") at the visit.
Time Frame: Week 6
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | NBI-98854 Low Dose | NBI-98854 High Dose
Number analyzed (Participants) | 29 | 30 | 31
Participants | 6 | 6 | 11
Statistical Analysis 1: Comparison: Placebo vs NBI-98854 High Dose; Test type: Superiority; p = 0.18, Cochran-Mantel-Haenszel — Comparison was not included in multiplicity adjustment procedure; Stratified by age group (6 to 11 years, 12 to 17 years); Risk Difference (RD) = 14.8 — Risk difference expressed as a percentage
Statistical Analysis 2: Comparison: Placebo vs NBI-98854 Low Dose; Test type: Superiority; p = 0.95, Cochran-Mantel-Haenszel — Comparison was not included in multiplicity adjustment procedure; Stratified by age group (6 to 11 years, 12 to 17 years); Risk Difference (RD) = -0.7 — Risk difference expressed as a percentage

ADVERSE EVENTS:
Time Frame: Up to 8 weeks
Description: Includes all participants who were randomized and dispensed study drug, with 2 exclusions: (a) participants who withdrew from study and returned all previously dispensed study drug with all doses present, and (b) participants who have no postbaseline safety data collected. Dose levels based on age group were prespecified to be combined within each dose arm.
Arm/Group | Placebo | NBI-98854 Low Dose | NBI-98854 High Dose
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/32 | 0/33
Serious Adverse Events (participants affected / at risk) | 1/32 | 0/32 | 0/33
Other Adverse Events (participants affected / at risk) | 9/32 | 15/32 | 19/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=32) | NBI-98854 Low Dose (N=32) | NBI-98854 High Dose (N=33)
Conversion disorder (Psychiatric disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=32) | NBI-98854 Low Dose (N=32) | NBI-98854 High Dose (N=33)
Headache (Nervous system disorders) | 3 | 6 | 3
Somnolence (Nervous system disorders) | 1 | 4 | 3
Sedation (Nervous system disorders) | 0 | 2 | 3
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 5
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 2
Sinusitis (Infections and infestations) | 0 | 0 | 2
Insomnia (Psychiatric disorders) | 1 | 2 | 3
Anxiety (Psychiatric disorders) | 1 | 0 | 2
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 2
Tic (Psychiatric disorders) | 2 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 2
Vomiting (Gastrointestinal disorders) | 1 | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 1
Irritability (General disorders) | 3 | 2 | 2
Fatigue (General disorders) | 0 | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Neutrophil count decreased (Investigations) | 0 | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Generally, the PI has the right to publish results provided such publication does not violate confidentiality or IP provisions within the contract with the Sponsor. Prior to submission for publication or presentation of results, the PI must provide the Sponsor time for review. The Sponsor can request the PI to withhold or remove information from all publications. For a multi-center study, any publication of results by the PI shall not be made before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2016-06-29): https://cdn.clinicaltrials.gov/large-docs/79/NCT02679079/Prot_000.pdf
  • Statistical Analysis Plan (2017-05-05): https://cdn.clinicaltrials.gov/large-docs/79/NCT02679079/SAP_001.pdf